CLINICAL TRIAL: NCT04069806
Title: An Analysis of Risk Factors and Implementation of Strategies to Prevent Nausea and Vomiting in Patients Undergoing Regional Anesthesia for Caesarean Section
Brief Title: Preoperative Oral Carbohydrate for Nausea and Vomiting Prevention During Cesarian Section
Acronym: POC-NaVoP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Katarzyna Kotfis, Primary Investigator, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PUM_08.08.2019
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Nausea; Vomiting; Oral carbohydrate; Fasting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting; Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative oral carbohydrate load (Experimental): 6 hours for solid food and 2 hours for liquids + oral carbohydrate preparation 2 hours prior to surgery.
  Interventions: Dietary Supplement: preoperative oral carbohydrate, preOp
- Standard preoperative fasting (No Intervention): 6 hours for solid food and 2 hours for liquids.

INTERVENTIONS:
Dietary Supplement: preoperative oral carbohydrate, preOp — Patients in the experimental arm will receive oral carbohydrate preparation at 2 hours prior to planned caesarian section.
  Arms: Preoperative oral carbohydrate load

SUMMARY:
Post-operative nausea and vomiting (PONV) in women undergoing subarachnoid anesthesia for Caesarean section is an important clinical problem. The aim of this study is to compare the effectiveness of oral carbohydrate loading to standard pre-operative fasting in patients undergoing elective cesarean section on the incidence and severity of PONV and biochemical parameters indicating ketosis.

DETAILED DESCRIPTION:
Post-operative nausea and vomiting (PONV) in women undergoing subarachnoid anesthesia for Caesarean section is an important clinical problem. Known mechanisms underlying PONV are based on prolonged fasting, hypotension due to concomitant sympatholysis during anesthesia, bradycardia due to increased vagal tone, visceral stimulation during surgery and intrathecal administered opioids. However, the identification of patients exposed to this problem and appropriate perioperative preparation is of key importance. An analysis of risk factors for postoperative nausea and vomiting in patients undergoing elective cesarean section under spinal anesthesia is of major clinical importance. The aim of this study is a comparison of the effectiveness of oral carbohydrate loading strategy as compared with standard pre-operative fasting in patients undergoing elective cesarean section under spinal anesthesia on the incidence and severity of PONV and biochemical parameters indicating ketosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years.
2. Scheduled for an elective cesarean section.
3. Uncomplicated pregnancy.
4. Planned for spinal anesthesia.
5. ASA I or ASA II.

Exclusion Criteria:

1. History of diabetes.
2. History of gastro-intestinal reflux (GERD).
3. Unable or unwilling to sign an informed consent.
4. Contraindications to spinal anesthesia.
5. Contraindication to Oral carbohydrate formula.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant patients scheduled for planned cesarian section.
Enrollment: 140 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting 6 hours after caesarian section. | 6 hours
  The Postoperative Nausea and Vomiting (PONV) Intensity Scale 6 hours after caesarian section. Scale range: 0-50. The scale measures PONV intensity, where a score ≥50 defined clinically important PONV: PONV Intensity Scale=severity of nausea (1=mild, 2=moderate, 3=severe)×pattern of nausea (1=varying, 2=constant)×duration of nausea (in hours).
Postoperative nausea and vomiting 24 hours after caesarian section. | 24 hours
  The Postoperative Nausea and Vomiting (PONV) Intensity Scale 24 hours after caesarian section. Scale range: 0-50. The scale measures PONV intensity, where a score ≥50 defined clinically important PONV: PONV Intensity Scale=severity of nausea (1=mild, 2=moderate, 3=severe)×pattern of nausea (1=varying, 2=constant)×duration of nausea (in hours).

SECONDARY OUTCOMES:
Time to first peristalsis. | 24 hours
  Moment of first peristalsis after operation (in hours).
Time to first bowel movement. | 24 hours
  Moment of first bowel movement after operation (in hours).
Concentration of serum lactate in serum. | 0 hours
  Lactate level measured in maternal serum.
Concentration of beta-hydroxy-butiric acid in serum. | 0 hours
  Beta-hydroxy-butiric acid level measured in maternal serum.
Insulin resistance factor (HOMA-IR). | 0 hours
  Insulin resistance measured in maternal serum.
Concentration of isoprostane in urine. | 0 hours
  Isoprostane level measured in maternal urine.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna L Kotfis, MD, PhD, Principal Investigator — Pomeranian Medical University; Sebastian Kwiatkowski, MD, PhD, Study Chair — Pomeranian Medical University
Locations (1):
- Pomeranian Medical University, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kotfis K, Jamiol-Milc D, Wojciechowska A, Szylinska A, Drozd A, Zimny M, Dolegowska B, Kwiatkowski S, Dziedziejko V, Safranow K. Maternal and umbilical cord plasma purine concentrations after oral carbohydrate loading prior to elective Cesarean delivery under spinal anesthesia: a randomized controlled trial. BMC Pregnancy Childbirth. 2025 May 10;25(1):556. doi: 10.1186/s12884-025-07637-6. PMID 40348958
- [Derived] Kotfis K, Wojciechowska A, Zimny M, Jamiol-Milc D, Szylinska A, Kwiatkowski S, Kaim K, Dolegowska B, Stachowska E, Zukowski M, Pankowiak M, Torbe A, Wischmeyer P. Preoperative Oral Carbohydrate (CHO) Supplementation Is Beneficial for Clinical and Biochemical Outcomes in Patients Undergoing Elective Cesarean Delivery under Spinal Anaesthesia-A Randomized Controlled Trial. J Clin Med. 2023 Jul 28;12(15):4978. doi: 10.3390/jcm12154978. PMID 37568381